CLINICAL TRIAL: NCT02307058
Title: A Phase II Randomized Trial of MRI-Guided Prostate Boosts Via Initial Lattice Stereotactic vs Daily Moderately Hypofractionated Radiotherapy - The Miami BLaStM Trial
Brief Title: Randomized MRI-Guided Prostate Boosts Via Initial Lattice Stereotactic vs Daily Moderately Hypofractionated Radiotherapy
Acronym: BLaStM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Alan Pollack, MD, PhD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140627
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LEAD RT Group (Experimental): Participants in this group will receive the Lattice Extreme Ablative Dose (LEAD) radiotherapy. Radiotherapy will begin within two months of fiducial marker placement. The therapy will consist of 39 fractions over approximately 8 weeks.
  Interventions: Radiation: LEAD RT
- HEIGHT RT Group (Experimental): Participants in this group will receive the Hypofractionated Extended Image-Guided Highly Targeted (HEIGHT) radiotherapy. Radiotherapy will begin within two months of fiducial marker placement. The therapy will consist of 39 fractions over approximately 7 and a half weeks.
  Interventions: Radiation: HEIGHT RT

INTERVENTIONS:
Radiation: LEAD RT — The multiparametric-MRI (MP-MRI) defined Gross Tumor Volume (GTV) will receive 12-14 Gy on the first day of treatment and then the prostate plus proximal seminal vesicles (SV), the Clinical Target Volume (CTV)1, will receive 76 Gy in 38 fractions (Fxs) at 2.0 Gy per Fx. For High Risk patients, the distal SVs may be treated to 56 Gy in 38 Fxs or full dose (CTV2), and the pelvic lymph nodes may be treated to 56 Gy in 38 Fxs (CTV3).
  Other Names: Stereotactic Lattice Radiation Therapy
  Arms: LEAD RT Group
Radiation: HEIGHT RT — The MRI defined GTV(s) will receive a higher dose per day than the CTV by dose painting. The GTV(s) will receive an absolute dose of 91.2 Gy. Assuming an α/β ratio of 3.0, this would be equivalent to 98.5 Gy in 2.0 Gy fractions. The prostate plus proximal seminal vesicles (CTV1) will receive 76 Gy in 38 fractions (Fxs) at 2.0 Gy per Fx. For High Risk patients, the distal SVs (CTV2) may be treated to 56 Gy in 38 Fxs or full dose, and the pelvic lymph nodes (CTV3) may be treated to 56 Gy in 38 Fxs.
  Other Names: Moderate Hypofractionation Radiation Therapy
  Arms: HEIGHT RT Group

SUMMARY:
The purpose of this research study is to learn about: 1) improving control of prostate cancer using an extra high dose radiation treatment to the MRI defined high risk tumor areas, in addition to the standard radiation treatment to the rest of the prostate; 2) preserving quality of life by reducing dose to the nearby organs at risk around the prostate; and 3) establishing the relationship of pre- and post-treatment MRI to MRI-directed biopsy results at 2-2.5 years after treatment.

ELIGIBILITY:
Eligibility Criteria:

* A. Biopsy confirmed adenocarcinoma (including ductal) of the prostate.
* B. T1-T3 disease based on digital rectal exam.
* C. No evidence of metastasis by any clinical criteria or available radiographic tests (N0M0 by clinical or imaging criteria).
* D. Gleason score 6-10.
* E. Androgen deprivation therapy (ADT) is at the discretion of the treating physician; but, must be decided (none, short-term or long-term as counted from the luteinizing hormone-releasing hormone (LHRH) agonist or antagonist injection) prior to enrollment. An anti-androgen (e.g., bicalutamide at 50 mg per day po) is recommended to start prior to LHRH agonist injection (not recommended for LHRH antagonist injection) and is recommended to not be administered for more than 4 months. If ADT is planned, the following restrictions apply:

  * i. It may be initiated no more than 3 months prior to the signing of consent
  * ii. It must be started prior to the start of radiotherapy and
  * iii. The total length planned must be ≤ 30 months
* F. Prostate-specific Antigen (PSA) ≤ 100 ng/mL within (+/-) 4 months of signing of consent. If PSA was above 100 and drops to ≤ 100 with antibiotics, this is acceptable for enrollment.
* G. Subjects with T3 disease based on digital rectal exam (DRE), Gleason 8-10 or a PSA of >15 ng/ml, should have a bone scan within (+/-) 4 months of signing of consent that is without evidence of metastasis. A questionable bone scan is acceptable if additional imaging studies (e.g., plain x-rays, CT, or MRI) do not confirm for metastasis.
* H. Suspicious peripheral zone or central gland lesion on MP-MRI

  * i. Peripheral zone: Distinct lesion on dynamic contrast-enhanced MRI (DCE-MRI) with early enhancement and later washout (Note: contrast not required for enrollment), and/or distinct lesion on the ADC map (Value <1000).
  * ii. Central gland: A suspicious central gland lesion on MP-MRI must have a distinct lesion on the apparent diffusion coefficient (ADC) map (Value <1000)
* I. No previous pelvic radiotherapy.
* J. No previous history of radical/total prostatectomy (suprapubic prostatectomy is acceptable).
* K. No concurrent, active malignancy, other than nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for ≥ 5 years then the patient is eligible.
* L. Ability to understand and the willingness to sign a written informed consent document.
* M. Zubrod performance status ≤ 2. (Karnofsky or Eastern Cooperative Oncology Group (ECOG) performance status may be used to estimate Zubrod).
* N. Willingness to fill out quality of life/psychosocial forms.
* O. Age ≥ 35 and ≤ 85 years at signing of consent.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2015-02-05 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Early Prostate Tumor Response (EPTR) | Up to 3 years
  Prostate Tumor Pathologic Complete Response (PathCR measured using ultrasound guided systematic prostate biopsy) and/or early biochemical response at 9 months post-RT.

SECONDARY OUTCOMES:
Correlation between EPTR and Changes in serial post-RT MRIs | 3 months post-RT, 9-months post-RT, within 3 months of 2-2.5 post-treatment biopsy
  To establish the relationship between EPTR and changes in serial post-RT MRI's obtained at 3 months and 9 months after RT, and within 3 months prior to the primary endpoint post-treatment prostate biopsy at 2.0-2.5 yr after completion of all therapy.
Number of participants experiencing treatment related adverse events | Up to 2 years
  Number of participants experiencing acute and late toxicity will be evaluated by treating physicians
Health-Related Quality of Life Scores: EPIC SF-12 | Up to 5.25 years (post-treatment)
  Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite and Medical Outcomes Study SF-12 (EPIC SF-12) to evaluate patient function and satisfaction after prostate cancer treatment. Response options for each item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Health-Related Quality of Life Scores: MAX-PC | Up to 5.25 years (post-treatment)
  Health-related quality of life (HRQOL) will be measured using the scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer (MAX-PC) from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
Health-Related Quality of Life Scores: IPSS | Up to 5.25 years (post-treatment)
  Health-related quality of life (HRQOL) will be measured using the International Prostate Symptom Score (IPSS) to evaluate patient urinary function and quality of life. There are 7 questions related to urinary function. Responses are on a scale from 0 ("not at all") to 5 ("almost always"), with higher scores indicating higher levels of urinary dysfunction. There is 1 quality of life question related to urinary symptoms. Responses are on a scale from 0 ("delighted") to 6 ("terrible").
Change in gene/biomarker expression | Baseline, Up to 5.25 years (post-treatment)
  Change in gene/biomarker expression in different MP-MRI tumor regions assessed from prostate biopsy samples.
Rate of participant response | Up to 5.25 years (post-treatment)
  Participant response will be reported as the percentage of participants with reported biochemical failure (defined as having an increase of 2 ng/mL PSA levels from nadir), clinical failure (defined as having evidence of distant metastasis and overall failure), cause specific mortality and overall mortality.
Change in CTC Levels | Baseline (pre-treatment), Up to 2 years (post-treatment)
  Circulating Tumor Cell (CTC) levels evaluated from peripheral blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Some data after completion of the trial and publication of the primary endpoint. Additional data after publication of the secondary endpoints.